CLINICAL TRIAL: NCT06326177
Title: Investigating Association Between Spine Posture, Spine Movement, Scapular Dyskinesia, Isometric and Eccentric Shoulder Strength and Core Muscle Endurance in Competitive Swimmers
Brief Title: Investigating Association Between Spine, Scapular, Shoulder and Core in Swimmers
Status: Enrolling by invitation | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Poyraz Tuncer, Physiotherapist, Yeditepe University
Other Study IDs: Yeditepe U - Poyraz Tuncer
Record Dates: First submitted 2024-03-05; First posted 2024-03-22 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Postural Kyphosis; Postural Lordosis; Movement, Abnormal; Spine Injury; Cervical Lordosis
MeSH Terms: conditions — Dyskinesias; Spinal Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Competitive Swimmer Group: Spine posture, spine movement, scapular dyskinesia, ısometric and eccentric shoulder strength and core muscle endurance will be assessed.
  Interventions: Procedure: Spine Posture Assessment; Procedure: Spine Movement Assessment; Procedure: Core Muscle Endurance Assessment; Procedure: Scapular Dyskinesia; Procedure: Shoulder Strength
- Recreational Swimmer Group: Spine posture, spine movement, scapular dyskinesia, ısometric and eccentric shoulder strength and core muscle endurance will be assessed.
  Interventions: Procedure: Spine Posture Assessment; Procedure: Spine Movement Assessment; Procedure: Core Muscle Endurance Assessment; Procedure: Scapular Dyskinesia; Procedure: Shoulder Strength

INTERVENTIONS:
Procedure: Spine Posture Assessment — Spine posture will be assessed with double inclinometer method. After determining landmarks for each assessment, inclinometers will be placed and degree will be noted. Both degree which are obtained with different inclinometers will be used to summed up for determining postural alteration degree. Cervical, thoracal, thoracolumbar and lumbar spinal postures will be used. Spine postures are going to be expressed as, cervical lordosis degree, thoracal kyphosis degree, thoracolumbar posture degree and lumbar lordosis degree. Landmarks for cervical lordosis are C2 and C7, for thoracal kyphosis are T1 and T12, for lumbar lordosis are T12 and S1, for thoracolumbar posture C7 and S1.
Procedure: Spine Movement Assessment — Spine movement will be assessed via using bubble inclinometer in terms of degree. Bony landmarks will be spotted like done in spine posture assessment after that full spinal flexion and extension wanted in order to record degrees in inclinometers at the end range. As a result the difference between two inclinometer will give the motion of that segment. Lumbar and thoracolumbar spinal movement will be assessed with this method. For thoracal and cervical range of motion values will be recorded separately without substruction from both inclinometer. Thoracal rotation range of motion will be assessed with two landmarks and will be recorded separately according to landmark. Thoracolumbar range of motion will be assessed with two substruction of degrees. Landmarks for cervical range of motion are vertex and C7, for thoracal range of motion are T1 and T12, for lumbar range of motion are T12 and S1, for thoracolumbar range of motion C7 and S1.
Procedure: Core Muscle Endurance Assessment — Core muscle endurance is divided into three components. Trunk anterior flexion test will be used to assess anterior core region endurance. Lateral plank test will be used to determine lateral core muscle endurance. Trunk posterior extensor test will be used to determine endurance of the posterior core musculature. All of these test are calculated in predetermined positions according to literature with static contractions. Maximum duration of maintaining that position is needed. In trunk anterior flexion test participant will sit with 60 degree inclination from the ground while making contact with their feet when hips and knees are flexed. In lateral plank test participants should place their elbow to ground and lift their hip while feet are in contact with ground in side lying position. In trunk extensor endurance test participants will lie prone to the bed while maintaining contact with their ASIS and lower extremity. The upper body should stay outside of the bed.
Procedure: Scapular Dyskinesia — Scapular dyskinesia will be assessed with scapular dyskinesia test. Dumbbells which are 1,5kg will be used in the testing setting. Participant will perform full shoulder abduction for 5 times while examiner assesses the movement quality by ranking it as subtle dyskinesis, obvious dyskinesis and no dyskinesis according to the movement of the scapula. After that participant will perform 5 repetitions of shoulder flexion.
Procedure: Shoulder Strength — Shoulder strength will be assessed via usage of microfet hand held dynamometer. Isometric shoulder strength will be calculated in supine lying position while participant holding their arm at side with 90 degree elbow flexion. After that participant will apply maximal contraction towards external rotation while examiner resists that motion in order to prevent any motion with dynamometer. Eccentric shoulder strength will be assessed in sitting position. Participant will hold their shoulder at 90 degrees of abduction with 90 degree external rotation. Also elbow should be in 90 degree flexed position. After that examiner will give force towards neutral rotation while holding the arm. Participant will resist this motion eccentrically until neutral rotation is reached. Velocity of the shoulder should be same throughout all motion due to creation of isokinetic environment.

SUMMARY:
The aim of this observational study is to investigate relationship between cervical, thoracic, lumbar and thoracolumbar spine posture, spine movement, isometric and eccentric shoulder strength, scapular dyskinesis and core muscle endurance in healthy competitive young swimmers in comparison with healthy recreational swimmers. The main question is whether spine posture affects spine movement, shoulder strength, scapular dyskinesia and core endurance. Participants will asked to complete a warm up period, after that spine posture, spine movement, scapular dyskinesia, shoulder strength and core endurance will be assessed by examiner. Researchers will compare competitive swimmer group and recreational swimmer group. Additionally correlation between spine posture, spine movement, scapular dyskinesia, shoulder strength and core muscle endurance will be investigated in competitive swimmer group. Aim of the study is to determine whether posture have any effect upon these parameters.

DETAILED DESCRIPTION:
The aim of this observational study is to investigate relationship between cervical, thoracic, lumbar and thoracolumbar spine posture, spine movement, scapular dyskinesia, shoulder strength and core muscle endurance in healthy competitive youth swimmers in comparison with healthy recreational swimmers. Study expected to include 44 participants which is distributed into experiment (n=22) and control (n=22) groups. The participants will be taken from Turkish swimming clubs which are Fenerbahçe, Galatasaray, ENKA, etc. between march and may of 2024. All of the research will be done in PT Academy clinic which is located in Turkey. The ages of the swimmers will be between 12-24. Experiment group should be a competitive swimmer that were also, participating swimming training in 6 days a week which is consisting of at least 12 hours of swimming training. They should pass Turkish swimming championship qualification times in order to participate in this study. Participants who have any systemic, neurologic, tumoral and cardiopulmonary pathologies excluded. Swimmers that compete in open water races are excluded. Participants that had orthopedic problem or surgical procedure in the past 6 months had been excluded. Inclusion criteria of the control group are different than the experiment group. They don't need to be a competitive swimmer as well as they don't need prerequisites of being a competitive swimmer. But, exclusion criteria remained same with experimental group except being open water swimmer. Before assessments participants will perform 10 minutes of warm up consisting of thigh, arm and core muscles as well as steady state aerobic exercise. Cervical lordosis, thoracal kyphosis, lumbar lordosis and thoracolumbar position degree will be assessed with double inclinometer. Core endurance will be assessed with trunk anterior flexion test, trunk posterior extensor test and lateral plank test. Ratios of core endurance parameters will be used in statistical analysis in order to compare with normative data. Spinal movement will be assessed via bubble inclinometer. For spinal movement cervical, lumbar, thoracal and thoracolumbar flexion and extension motion will be assessed. Also, thoracal and thoracolumbar rotation range of motion will be recorded. Scapular dyskinesia test will be used in order to assess scapular dyskinesia. Shoulder strength will be assessed via using microfet hand held dynamometer. Both isometric and eccentric shoulder external rotation strength will be measured. Ratios between these two values will be used in the statistical analysis. Results will be compared with each other between competitive and recreational swimmer group. SPSS analysis system will be used in order to make statistical analysis. For mean analysis t test or Mann Whitney u test will be used according to distributions of the groups. For the correlation analysis regression and mediation analysis will be used. Mean comparison will be done in between group setting. On the other hand correlation investigation of parameters will be done within group setting only including competitive swimmer group. As a result difference between recreational and competitive swimmers will be revealed as well as association between posture and other variables will be revealed with correlation between parameters.

ELIGIBILITY:
Inclusion Criteria:

* Being a competitive swimmer.
* Being between 12-24 ages.
* Participating swimming training at least 6 days a week.
* Swimming faster than Turkish National Championship participation qualification times in their age group.
* Participating swimming training at least 12 hours a week.
* Should start swimming at least 6 years before.

Exclusion Criteria:

* Being an open water swimmer.
* Having systemic, cardiopulmonary and neurological pathology.
* Having orthopedic pathology in the past 6 months.
* Having surgical history in past 6 months.
* Having tumoral condition.
* Having spine pathology in past 6 months.

Inclusion criteria for control group:

* Being a recreational swimmer.
* Being between 12-24 ages.

Exclusion criteria for control group:

* Having systemic, cardiopulmonary and neurological pathology.
* Having orthopedic pathology in the past 6 months.
* Having surgical history in past 6 months.
* Having tumoral condition.
* Having spine pathology in past 6 months.

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Study population will be selected from swimmers in Fenerbahçe, Galatasaray, ENKA, İstek and TOHM clubs. Study takes place in İstanbul. Study will include swimmers that are also swimming in USA for their university teams due to their education which are also competing in Turkey for their aforementioned clubs in the Turkish Championship. Participant pool approximately between 200-300 swimmers. Both gender will be included.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2024-08-10 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Spinal Posture | 1 Day
  Cervical lordosis, thoracal kyphosis, lumbar lordosis and thoracolumbar posture will be recorded. All parameters will be calculated in degree.
Cervical Movement | 1 Day
  Cervical flexion and extension will be calculated. All parameters will be calculated in degree.
Thoracic Movement | 1 Day
  Thoracic flexion and extension will be recorded. Also thoracal rotation will be recorded. All parameters will be calculated in degree.
Lumbar Movement | 1 Day
  Lumbar flexion and extension will be recorded. All parameters will be calculated in degree.
Thoracolumbar Movement | 1 Day
  Thoracolumbar flexion and extension will be recorded. Thoracolumbar rotation will be recorded. All parameters will be calculated in degree.

SECONDARY OUTCOMES:
Anterior Core Musculature Assessment | 1 Day
  Trunk anterior flexion test will be used to assess anterior core region endurance. Score will be calculated in seconds.
Lateral Core Musculature Assessment | 1 Day
  Lateral plank test will be used to determine lateral core muscle endurance. Score will be calculated in seconds.
Posterior Core Musculature Assessment | 1 Day
  Trunk posterior extensor test will be used to determine endurance of the posterior core musculature. Score will be calculated in seconds.
Core Musculature Ratio Assessment | 1 Day
  Trunk anterior musculature and trunk posterior musculature ratio, ratio of two sides of lateral core musculature and lateral trunk musculature and extensor trunk musculature will be used.
Shoulder Strength Assessment | 1 Day
  Isometric and eccentric shoulder external rotation strength will be recorded in Newton unit.
Shoulder Strength Ratio Assessment | 1 Day
  Ratio between shoulder internal rotation and external rotation strength will be used.
Scapular Dyskinesia | 1 Day
  Scapular dyskinesia will be recorded with Scapular Dyskinesia Test by using dumbbells which was described by McClure. Scapular dyskinesia will be measure as normal scapular motion, subtle dyskinesis and obvious dyskinesis.

CONTACTS AND LOCATIONS:
Locations (1):
- PT Academy, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Only result and certain characteristics may be shared.

REFERENCES:
- [Background] Lewis JS, Wright C, Green A. Subacromial impingement syndrome: the effect of changing posture on shoulder range of movement. J Orthop Sports Phys Ther. 2005 Feb;35(2):72-87. doi: 10.2519/jospt.2005.35.2.72. PMID 15773565
- [Background] Dimitriadis Z, Parintas I, Karamitanis G, Abdelmesseh K, Koumantakis GA, Kastrinis A. Reliability and Validity of the Double Inclinometer Method for Assessing Thoracolumbar Joint Position Sense and Range of Movement in Patients with a Recent History of Low Back Pain. Healthcare (Basel). 2022 Dec 29;11(1):105. doi: 10.3390/healthcare11010105. PMID 36611565
- [Background] Abdelraouf OR, Abdel-Aziem AA. THE RELATIONSHIP BETWEEN CORE ENDURANCE AND BACK DYSFUNCTION IN COLLEGIATE MALE ATHLETES WITH AND WITHOUT NONSPECIFIC LOW BACK PAIN. Int J Sports Phys Ther. 2016 Jun;11(3):337-44. PMID 27274419
- [Background] Kolber MJ, Pizzini M, Robinson A, Yanez D, Hanney WJ. The reliability and concurrent validity of measurements used to quantify lumbar spine mobility: an analysis of an iphone(R) application and gravity based inclinometry. Int J Sports Phys Ther. 2013 Apr;8(2):129-37. PMID 23593551
- [Background] Salamh PA, Kolber M. The reliability, minimal detectable change and concurrent validity of a gravity-based bubble inclinometer and iphone application for measuring standing lumbar lordosis. Physiother Theory Pract. 2014 Jan;30(1):62-7. doi: 10.3109/09593985.2013.800174. Epub 2013 Jul 17. PMID 23862655
- [Background] Mayer TG, Tencer AF, Kristoferson S, Mooney V. Use of noninvasive techniques for quantification of spinal range-of-motion in normal subjects and chronic low-back dysfunction patients. Spine (Phila Pa 1976). 1984 Sep;9(6):588-95. doi: 10.1097/00007632-198409000-00009. PMID 6238424
- [Background] Laudner K, Lynall R, Williams JG, Wong R, Onuki T, Meister K. Thoracolumbar range of motion in baseball pitchers and position players. Int J Sports Phys Ther. 2013 Dec;8(6):777-83. PMID 24377063
- [Background] van Baalen GB, Vanwanseele B, Venter RR. Reliability and Validity of a Smartphone Device and Clinical Tools for Thoracic Spine Mobility Assessments. Sensors (Basel). 2023 Sep 2;23(17):7622. doi: 10.3390/s23177622. PMID 37688076
- [Background] Holt KL, Raper DP, Boettcher CE, Waddington GS, Drew MK. Hand-held dynamometry strength measures for internal and external rotation demonstrate superior reliability, lower minimal detectable change and higher correlation to isokinetic dynamometry than externally-fixed dynamometry of the shoulder. Phys Ther Sport. 2016 Sep;21:75-81. doi: 10.1016/j.ptsp.2016.07.001. Epub 2016 Jul 9. PMID 27500450
- [Background] Johansson FR, Skillgate E, Lapauw ML, Clijmans D, Deneulin VP, Palmans T, Engineer HK, Cools AM. Measuring Eccentric Strength of the Shoulder External Rotators Using a Handheld Dynamometer: Reliability and Validity. J Athl Train. 2015 Jul;50(7):719-25. doi: 10.4085/1062-6050-49.3.72. Epub 2015 May 14. PMID 25974381
- [Background] Uga D, Endo Y, Nakazawa R, Sakamoto M. Electromyographic analysis of the infraspinatus and scapular stabilizing muscles during isometric shoulder external rotation at various shoulder elevation angles. J Phys Ther Sci. 2016 Jan;28(1):154-8. doi: 10.1589/jpts.28.154. Epub 2016 Jan 30. PMID 26957748
- [Background] Papotto BM, Rice T, Malone T, Butterfield T, Uhl TL. Reliability of Isometric and Eccentric Isokinetic Shoulder External Rotation. J Sport Rehabil. 2016 Jun 6;25(2):2015-0046. doi: 10.1123/jsr.2015-0046. Print 2016 May 1. PMID 26562351
- [Background] Tate AR, McClure P, Kareha S, Irwin D, Barbe MF. A clinical method for identifying scapular dyskinesis, part 2: validity. J Athl Train. 2009 Mar-Apr;44(2):165-73. doi: 10.4085/1062-6050-44.2.165. PMID 19295961
- [Background] McClure P, Tate AR, Kareha S, Irwin D, Zlupko E. A clinical method for identifying scapular dyskinesis, part 1: reliability. J Athl Train. 2009 Mar-Apr;44(2):160-4. doi: 10.4085/1062-6050-44.2.160. PMID 19295960
- [Background] McFarland C, Wang-Price S, Richard S. Clinical measurements of cervical lordosis using flexirule and inclinometer methods in individuals with and without cervical spine dysfunction: A reliability and validity study. J Back Musculoskelet Rehabil. 2015;28(2):295-302. doi: 10.3233/BMR-140517. PMID 25096317
- [Background] Tawde P, Dabadghav R, Bedekar N, Shyam A, Sancheti P. Assessment of cervical range of motion, cervical core strength and scapular dyskinesia in violin players. Int J Occup Saf Ergon. 2016 Dec;22(4):572-576. doi: 10.1080/10803548.2016.1181892. Epub 2016 May 27. PMID 27232160
- [Background] Wolfenberger VA, Bui Q, Batenchuk GB. A comparison of methods of evaluating cervical range of motion. J Manipulative Physiol Ther. 2002 Mar-Apr;25(3):154-60. doi: 10.1067/mmt.2002.122327. PMID 11986576